CLINICAL TRIAL: NCT03819335
Title: ¿Puede Una aplicación móvil Mejorar el Conocimiento y la autogestión de Las Personas Con Diabetes Tipo 1? Evaluación clínica de la App mySugr
Brief Title: ¿Can mySugr App Improve Knowledge and Self-management of People With Type 1 Diabetes Mellitus?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIBSP-SUG-2018-01
Record Dates: First submitted 2019-01-22; First posted 2019-01-28 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Mobile Applications; Telemedicine
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Active Comparator): Usual follow-up of diabetes type 1 with face-to-face visits
  Interventions: Other: Standard care
- mySugr app (Experimental): Telemedical assistance with mySugr app
  Interventions: Device: mySugr app

INTERVENTIONS:
Device: mySugr app — mySugr is a mobile medical app for diabetes management. It has been developed by Roche Diabetes Care and it has two versions, free and Pro. It allows to carry out the diary of diabetes, including the collection and analysis of data on glycaemia, food, physical activity or insulin dose. In addition, it is compatible with continuous glucose measurement systems. It has the possibility to add functionalities such as estimation of HbA1c levels, more detailed data analysis or integration with Google Fit type motion sensors, as well as a bolus calculator, reminders for measuring blood glucose or photo gallery in the Pro version, which is the one that will be provided to the patients for the study.
  Arms: mySugr app
Other: Standard care — Face-to-face visits
  Arms: Standard care

SUMMARY:
This project is based on the contribution that an app can offer for improving knowledge and self-management of people with type 1 diabetes.

The main objective of this study is to assess mySugr app as a tool for empowering people with type 1 diabetes.

The study population are type 1 diabetes people, aged more than 18 years old and with more than one year from diagnosis. They will be randomised to standard care or use of mySugr app and will be followed-up during 48 weeks.

Control group will attend 5 face-to-face visits (baseline, 3, 6, 9 and 12 months) with the possibility of telephone contact and hospital assistance if necessary. Intervention group will attend 3 face-to-face visits (baseline, 6 and 12 months) and 2 telematic visits (at 3 and 9 months) and will also have the possibility of telephone contact and hospital assistance if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* People with type 1 diabetes (> 1 year diagnosis)
* Treatment with insulin in basal-bolus regimen
* Glucometer that connects automatically with the app
* HbA1c 7-9%
* Understanding of carbohydrate counting and concepts of ratio and factor of sensitivity
* Have a smartphone or tablet

Exclusion Criteria:

* Use at the time of randomization of another app for diabetes management
* Use of continuous monitoring or flash glucose systems
* Pregnancy
* Any other disease or condition that may interfere with the completion of the protocol or completion of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Empowerment | Baseline visit and month 12
  Change from baseline score in the Diabetes Empowerment Scale-Short Form Spanish version (DES-SF-S) (8, worse to 40, better) at 12 months

SECONDARY OUTCOMES:
Adherence to glycemic monitoring | Baseline visit and month 3, 6, 9 and 12
  Change from baseline frequency of glycemic monitoring (number of capillary blood glucose tests per day) at each follow-up visit
Adherence to recommendations | Each follow-up visit (month 3, 6, 9 and 12)
  Percentage of recommendations given by the medical team followed
Adherence to visits | Each follow-up visit (month 3, 6, 9 and 12)
  Percentage of face-to-face visits and telematic visits attended
Adherence to the app | End of the study (month 12) and 3 months after
  Percentage of patients who continue using the app after the end of the study
Daily management of diabetes | Baseline visit and month 12
  Change from baseline score in the questionnaire that evaluates the number of tasks performed in relation to diabetes (ad hoc) at 12 months
Quality of life related to diabetes | Baseline visit and month 12
  Change from baseline score in the Spanish version of the Diabetes Quality Of Life questionnaire (EsDQOL) (satisfaction: 75, worse, to 15, better; impact: 85, worse, to 17, better; social and vocational concern: 45, worse, to 7, better; concern related to diabetes: 20, worse, to 4, better) at 12 months
Self-efficacy | Baseline visit and month 12
  Change from baseline score in the Diabetes Distress Scale Spanish version (DSS-S) (102, worse, to 17, better) at 12 months
Glycemic control | Baseline visit and month 3, 6, 9 and 12
  Change from baseline mean blood glucose (mg/dl), standard deviation, low and high blood glucose index at each follow-up visit
Glycemic control | Baseline visit and month 6 and 12
  Change from baseline HbA1c DCA (%) at 6 and 12 months
Satisfaction with the app | End of the study (month 12)
  Score in the satisfaction questionnaire in relation to the use of the platform (ad hoc)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cuixart G, Corcoy R, Gonzalez C. Can a mobile application improve glucose-related and patient-reported outcome measures (PROMs) in people with type 1 diabetes mellitus? A randomized controlled trial using the mySugr(R) app. Hormones (Athens). 2025 Mar;24(1):137-147. doi: 10.1007/s42000-024-00609-z. Epub 2024 Oct 16. PMID 39412732